CLINICAL TRIAL: NCT02835911
Title: LCCC 1229: Developing a Prospective Lymphoma Clinical Cohort in Malawi
Brief Title: Clinical Cohort of Lymphoma Patients in Malawi
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 1229; K01TW009488 (NIH)
Record Dates: First submitted 2016-01-19; First posted 2016-07-18 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Hematologic Malignancies
MeSH Terms: conditions — Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Left-over blood and tissue to be stored for future research testing.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lymphoma: Suspected lymphoma with confirmed hematologic malignancies treated under local conditions

SUMMARY:
This registry study is intended to establish a large prospective longitudinal clinical cohort of lymphoma patients in Malawi, as such data is currently lacking from sub-Saharan Africa. The investigators will perform core biopsies on at least 800 consecutively enrolled patients with suspected lymphoma for accurate histopathologic characterization. The investigators will systematically collect relevant clinical and laboratory data, and longitudinally follow those with confirmed hematologic malignancies receiving treatment according to local standards of care to assess outcomes.

DETAILED DESCRIPTION:
This is an observational cohort registry study of at least 800 patients with suspected lymphoma in Malawi. The primary purpose of this study is to develop a large prospective longitudinal lymphoma cohort at Kamuzu Central Hospital (KCH). Subjects with confirmed hematologic malignancies treated according to local standards of care will be actively followed for 2 years after diagnosis to assess clinical outcomes. After 2 years, if subjects are well, they will be discharged from clinic if they desire and contacted via telephone every 6 months for 5 years after lymphoma diagnosis simply to assess vital status. Subjects who wish to continue clinic follow-up after 2 years will be seen every 6 months until 5 years after lymphoma diagnosis. Those who are unwell after 2 years and continuing to receive active treatment will continue follow-up in clinic with all treatment details recorded.

All study laboratories and procedures which are being performed are consistent with international standards of care. Even without study implementation, all procedures may be undergone by patients at KCH, and there is no 'new' intervention being provided by the study which is currently absent in Malawi. However, current clinical and laboratory assessments of lymphoma patients at KCH over time are typically highly inconsistent and incomplete by international standards, as a result of extreme scarcity of resources and personnel. It is therefore hoped that the study will provide greater standardization and uniformity in the longitudinal characterization of patients with lymphoma at KCH, and allow data collected to be used for clinical as well as research purposes, as such data from sub-Saharan Africa are lacking and can be tremendously informative.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Referred to Kamuzu Central Hospital (KCH) with clinically suspected lymphoma based on clinical impression of referring providers Age >5 years, or ≤5 years only if lymphoma has already been pathologically confirmed.
* No prior or concurrent histologically confirmed cancer diagnosis or receipt of cancer treatment.
* Residence <200 kilometers from KCH. Able to understand and comply with study procedures for the entire length of the study, with assistance of parent or guardian as applicable.
* Subject (or parent or guardian as applicable) able to understand and provide written consent in English or Chichewa.
* Informed consent reviewed and signed by patient, or for pediatric patients, from parent or guardian.

Exclusion Criteria:

* There are no exclusion criteria other than failure to meet inclusion criteria listed above.
* Patients may consent to participation in the study but refuse directed genomic analysis of their lymphoma specimens.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 800 patients with suspected lymphoma in Malawi.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2012-11; Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with suspected lymphoma | 5 years
  At the time of initial assessment, all patients will undergo diagnostic lymph node biopsy.

SECONDARY OUTCOMES:
Number of patients with Epstein-Barr virus (EBV) | 5 years
  Core biopsy specimens will be tested for the presence of EBV and extra serum sample at enrollment, mid-treatment, treatment completion, and 6 months to allow EBV viral load
Information collected on Clinical & HR Quality of Life Questionnaire | 5 years
  Clinical & HRQOL assessment
Number of patients with Kaposi's sarcoma-associated herpesvirus (KSHV) | 5 years
  Core biopsy specimens will be tested for the presence of KSHV and extra serum sample at enrollment, mid-treatment, treatment completion, and 6 months to allow EBV viral load
Number of B-Cell Lymphomas | 5 years
  Diagnostic lymph node biopsy
Number of patients with childhood Burkitt lymphoma (BL) | 5 years
  enrolling children ≤5 years with already pathologically confirmed BL diagnoses
Number of Non-Hodgkin lymphoma (NHL) | 5 years
  At the time of initial assessment, all patients will undergo diagnostic lymph node biopsy.
Number of patients with Non- Malignant disorders | 5 years
  At the time of initial assessment, all patients will undergo diagnostic lymph node biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Satish Gopal, MD, Principal Investigator — UNC-CH
Locations (1):
- UNC Project, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gondwe Y, Kudowa E, Tomoka T, Kasonkanji ED, Kaimila B, Zuze T, Mumba N, Kimani S, Mulenga M, Chimzimu F, Kampani C, Randall C, Lilly A, Gopal S, Fedoriw Y, Painschab M. Comparison of baseline lymphoma and HIV characteristics in Malawi before and after implementation of universal antiretroviral therapy. PLoS One. 2022 Sep 1;17(9):e0273408. doi: 10.1371/journal.pone.0273408. eCollection 2022. PMID 36048901
- [Derived] Kaimila B, van der Gronde T, Stanley C, Kasonkanji E, Chikasema M, Tewete B, Fox P, Gopal S. Salvage chemotherapy for adults with relapsed or refractory lymphoma in Malawi. Infect Agent Cancer. 2017 Aug 9;12:45. doi: 10.1186/s13027-017-0156-3. eCollection 2017. PMID 28808480
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org